CLINICAL TRIAL: NCT02541331
Title: Influence of Polyvalent Mechanical Bacterial Lysate ISMIGEN® on Clinical Course of Asthma and Related Immunological Parameters in Asthmatic Children (EOLIA Study): Randomised Double-blind Placebo-controlled Multicentre Parallel-group Study
Brief Title: Efficacy Of Bacterial Lysate In Asthmatic Children
Acronym: EOLIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lallemand Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LPI-1201
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Allergic Asthma
Keywords: IgE-dependent asthma
MeSH Terms: interventions — Broncho-Vaxom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ISMIGEN (Experimental): Treatment over 3 successive months with one daily tablet over 10 days followed by 20 days of rest
  Interventions: Biological: ISMIGEN
- PLACEBO (Placebo Comparator): Treatment over 3 successive months with one daily tablet over 10 days followed by 20 days of rest
  Interventions: Biological: PLACEBO

INTERVENTIONS:
Biological: ISMIGEN — Tablets of 30 billion organisms/mg - Sublingual use 1 tablet per day over 10 days for 3 successive months.
  Other Names: Polyvalent Mechanical Bacterial Lysate - PMBL
  Arms: ISMIGEN
Biological: PLACEBO — Matched tablets without any active substance.
  Arms: PLACEBO

SUMMARY:
This study evaluate the efficacy of Mechanical Bacterial Lysate (PMBL - Ismigen®) to improve the asthma control level (ACT score) as add-on treatment to routine asthma treatment in children aged 6 to 16 with uncontrolled or partly controlled asthma. Half of the 150 participants will receive Ismigen® and their current asthma therapy while the other half will receive Placebo and their current asthma treatment.

DETAILED DESCRIPTION:
Acute and recurrent respiratory infections of the upper and middle respiratory tracts in the paediatric population of asthmatic patients represent a leading clinical burden, particularly during the winter. Respiratory tract infections, mainly viral infection are important factors that exacerbate asthma course in children. Currently no clinical data demonstrated the benefit of oral or sublingual bacterial lysates on asthma clinical course in children apart from one trial with OM-85 BV (Bronchovaxom®) suggesting reduced number and duration of infection-related wheezing attacks in children with asthma wheezing.

Therefore it was hypothesized that PMBL (Ismigen®) used in asthmatic children should significantly improve asthma course and control. A seasonal approach of active prevention, based on full-fledged antibacterial oral vaccination would be useful to show the potential benefit of this type of products.

The Primary objective was to assess the benefit of Ismigen® versus Placebo on the mean ACT score after administration of a Polyvalent Mechanical Bacterial Lysate (PMBL - Ismigen®) as add-on to routine asthma treatment.

Secondary objectives investigated:

* the potential reduction (vs Placebo) of number of asthma exacerbations, time to first event with Ismigen®;
* the potential decrease in number of respiratory tract infections during the observation period (3-month treatment and 6-month follow-up) after treatment;
* the specific changes occurring in a panel of immunological markers as the result of Ismigen® effect (subset of 48 patients).

ELIGIBILITY:
Inclusion Criteria:

1. Children of both genders aged 6 to 16 years.
2. Allergic asthma diagnosis with at least one perennial allergen according to the Global Strategy for Asthma Management and Prevention (GINA 2012 guidelines) prior to screening visit.
3. Patient shows clinical characteristics of partly controlled or uncontrolled asthma according to GINA 2012.
4. Already treated with SABA prn and ICS or ICS + LABA during the previous 3 months.
5. Patient shows antigen-specific IgE against HDM ≥ class 2 or positive skin prick test or RAST for at least one perennial allergen.
6. Patient who had at least 2 exacerbations of asthma within the 12-mo period before V1.
7. Patient not treated with Polyvalent Mechanical Bacterial Lysate (Ismigen®) within the previous 6 months prior to Visit 1.

Exclusion Criteria:

1. Patient received mechanical or any other bacterial lysate immunostimulation within the previous 6 months before Visit 1.
2. Patient received oral/subcutaneous allergen-immunotherapy within the previous 6 months before Visit 1.
3. History of near fatal asthma (e.g. brittle asthma, hospitalization for asthma exacerbation in Intensive Care Unit).
4. Pregnant or breastfeeding woman.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in asthma control level (mean ACT or P-ACT) score | at 3-months
  The main criterion is the improvement in mean ACT/P-ACT score versus baseline (between-groups comparison)

SECONDARY OUTCOMES:
Time-dependent change in asthma control level (mean ACT or P-ACT) score | at 6-months and at 9-months
  Improvement in ACT/P-ACT score versus baseline (between-groups comparison)
Number of respiratory infections occurring during the 3-mo treatment and the 6-mo follow-up after treatment | at 3-months, at 6-months and at 9-months
  Comparison of frequency of events between groups during the observation period.
Time to first mild or severe asthma exacerbation | From baseline
  To assess the exacerbation-free time after baseline (between-groups comparison)
Standardized mean daily dose of Inhaled Corticosteroids (ICS) used | From baseline, up to the 9-month time point
  To assess the amount of current asthma treatment (ICS) required to maintain a stable asthma control level (between-groups comparison)
Frequency of short acting beta-2 agonists use as rescue medication | From baseline, up to the 9-month time point
  To assess the necessary amount of rescue medication to cure exacerbations (between-groups comparison)
Serum Immunoglobulins | At baseline and at 3-months
  Levels of total IgE, IgA, IgM, IgG (including IgG1, IgG2, IgG3, IgG4) (between-groups comparison, biology subset)
Serum antibacterial antibodies concentration | At baseline, at 3-weeks and at 3-months
  Specific immunological response to Ismigen vaccination: IgG levels of Streptococcus pneumonia, Haemophilus Influenzae, Staphylococcus aureus, Klebsiella pneumonia, Streptococcus pyogenes, Klebsiella Ozenae, Streptococcus group A-G (between-groups comparison, biology subset)
Blood Specific markers of Lymphocyte activation | At baseline and at 3-months
  Levels of CD23 (B cells), CD25 (T cells) and CD69 (T, B and NK cells) (between-groups comparison, biology subset)
Activation of CD4 T cells in peripheral blood | At baseline and at 3-months
  Flow cytometric analyses of Foxp3 and CD25 expression as markers of conversion of T cells into nTreg and iTreg (between-groups comparison, biology subset)
Specific T cells responses in peripheral blood mononuclear cells (PBMC) | At baseline, at 3-weeks and at 3-months
  Number of vaccine specific T cells positive to IFN-gamma, IL-4, IL-13 assessed as spot-forming units by ELISPOT assay (between-groups comparison, biology subset)
PAQLQ (Paediatric Asthma Quality of Life Questionnaire) and PACQLQ (Paediatric Asthma Caregivers Quality of Life Questionnaire) | At baseline and at 9-months
  Patient and caregiver auto-questionnaires to assess the change in quality of life relative to asthma (between-groups comparison)
Cumulative number of days with respiratory tract infections | From baseline, up to the 9-month time point
  Cumulative number of days with an event (Between-groups comparison)
Number of lost school days due to respiratory infections and to asthma exacerbations | From baseline, up to the 9-month time point
  Cumulative number of days of absences (Between-groups comparison)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Durmont, MD, Study Director — Lallemand Pharma International AG
Locations (4):
- Poland (4):
  - LASERMED Diagnosis and Treatment Centre, Chełm
  - Children University Hospital - Pneumology and Rheumatology Dept, Lublin
  - ALERGOTEST s.c. Medical Centre, Lublin
  - Medical Centre Lucyna and Andrzej Dymek, Zawadzkie

REFERENCES:
- [Background] Razi CH, Harmanci K, Abaci A, Ozdemir O, Hizli S, Renda R, Keskin F. The immunostimulant OM-85 BV prevents wheezing attacks in preschool children. J Allergy Clin Immunol. 2010 Oct;126(4):763-9. doi: 10.1016/j.jaci.2010.07.038. PMID 20920766
- [Background] Sly PD, Boner AL, Bjorksten B, Bush A, Custovic A, Eigenmann PA, Gern JE, Gerritsen J, Hamelmann E, Helms PJ, Lemanske RF, Martinez F, Pedersen S, Renz H, Sampson H, von Mutius E, Wahn U, Holt PG. Early identification of atopy in the prediction of persistent asthma in children. Lancet. 2008 Sep 20;372(9643):1100-6. doi: 10.1016/S0140-6736(08)61451-8. PMID 18805338
- [Background] Jackson DJ, Gangnon RE, Evans MD, Roberg KA, Anderson EL, Pappas TE, Printz MC, Lee WM, Shult PA, Reisdorf E, Carlson-Dakes KT, Salazar LP, DaSilva DF, Tisler CJ, Gern JE, Lemanske RF Jr. Wheezing rhinovirus illnesses in early life predict asthma development in high-risk children. Am J Respir Crit Care Med. 2008 Oct 1;178(7):667-72. doi: 10.1164/rccm.200802-309OC. Epub 2008 Jun 19. PMID 18565953
- [Derived] Bartkowiak-Emeryk M, Emeryk A, Rolinski J, Wawryk-Gawda E, Markut-Miotla E. Impact of Polyvalent Mechanical Bacterial Lysate on lymphocyte number and activity in asthmatic children: a randomized controlled trial. Allergy Asthma Clin Immunol. 2021 Jan 20;17(1):10. doi: 10.1186/s13223-020-00503-4. PMID 33472687
- [Derived] Emeryk A, Bartkowiak-Emeryk M, Raus Z, Braido F, Ferlazzo G, Melioli G. Mechanical bacterial lysate administration prevents exacerbation in allergic asthmatic children-The EOLIA study. Pediatr Allergy Immunol. 2018 Jun;29(4):394-401. doi: 10.1111/pai.12894. PMID 29575037